CLINICAL TRIAL: NCT02061436
Title: Multicenter Registry of Chronic Total Occlusion Interventions
Brief Title: Prospective Global Registry for the Study of Chronic Total Occlusion Intervention
Acronym: PROGRESS-CTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: #11-099
Record Dates: First submitted 2014-01-28; First posted 2014-02-12 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: chronic total occlusion, percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous coronary intervention (PCI) of chronic total occlusions (CTOs) is increasingly being performed in patients with advanced coronary artery disease, but there is limited information on the techniques utilized and the procedural outcomes. The goal of this multicenter, investigator initiated registry is to collect information on treatment strategies and outcomes of consecutive patients undergoing CTO PCI among various participating centers. The information collected will be used to determine the frequency of CTO PCI performed at the participating sites and examine the procedural strategies utilized, and the procedural (both immediate and during follow-up) outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CTO PCI at each of the participating centers.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing CTO PCI at each of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
procedural success of chronic total occlusion PCI | discharge from the hospital after PCI, which usually happens the day after the procedure
  Procedural success is defined as achievement of technical success with no in-hospital major adverse cardiac events (MACE). In-hospital MACE includes any of the following adverse events prior to hospital discharge: death from any cause, Q-wave myocardial infarction, urgent repeat target vessel revascularization with PCI or coronary bypass surgery, tamponade requiring pericardiocentesis or surgery, or stroke.

SECONDARY OUTCOMES:
technical success of chronic total occlusion PCI | discharge from the hospital after PCI, which usually happens the day after the procedure
  Technical success of CTO PCI was defined as successful CTO revascularization with achievement of <30% residual diameter stenosis within the treated segment and restoration of TIMI grade 3 antegrade flow.
major adverse cardiovascular events | discharge from the hospital after PCI (which usually happens the day after the procedure) and during clinically-indicated follow-up. There are no pre-specified follow-up time periods - patients are assessed if and when they come to receive clinical care.
  In-hospital major adverse cardiovascular events (MACE) include any of the following adverse events prior to hospital discharge: death from any cause, Q-wave myocardial infarction, urgent repeat target vessel revascularization with PCI or coronary bypass surgery, tamponade requiring pericardiocentesis or surgery, or stroke.
  MACE during clinical follow-up include death, myocardial infarction, target lesion and target vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (48):
- United States (42):
  - Banner Samaritan Health Center, Phoenix, Arizona
  - Little Rock VA Medical Center, Little Rock, Arkansas
  - San Diego VAMC and University of California, San Diego, California
  - Torrance Memorial Medical Center, Torrance, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Memorial Hospital, Jacksonville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital- Emory Heart and Vascular Center, Atlanta, Georgia
  - Wellstar Health System, Marietta, Georgia
  - Northwestern Bluhm Cardiovascular Institute, Chicago, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Tulane University Heart and Vascular Institute, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Minneapolis VA Healthcare System and University of Minnesota, Minneapolis, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - Maimonides Medical Center, Brooklyn, New York
  - Trinity Medical WNY, Buffalo, New York
  - Columbia University, New York, New York
  - Carolina East Medical Center, New Bern, North Carolina
  - The Christ Hospital Ohio Heart & Vascular, Cincinnati, Ohio
  - University Hospitals (UH) Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Kettering Health Network, Kettering, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Hillcrest Medical Center, Tulsa, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - University of Pittsburgh Medical Center Presbyterian, Pittsburgh, Pennsylvania
  - WellSpan Heart & Vascular, York, Pennsylvania
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - VA Dallas Medical Center, Dallas, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White Research Institute-The Heart Hospital Baylor Plano, Plano, Texas
  - Baylor Scott and White Research Institute/ The Heart Hospital Baylor Plano, Plano, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Providence Health Center, Waco, Texas
  - Peacehealth Cardiology, Bellingham, Washington
  - Appleton Cardiology, Appleton, Wisconsin
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada
- Aswan Heart Centre, Aswān, Egypt
- Greece (2):
  - Korgialeneio-Benakeio Hellenic Red Cross General Hospital of Athens, Athens, Attica
  - Henry Hunant Hospital Center, Athens
- St. George Hospital University Medical Center, Beirut, Lebanon
- Meshalkin Novosibirsk Research Institute, Novosibirsk, Novosibirsk Oblast, Russia

REFERENCES:
- [Result] Christopoulos G, Menon RV, Karmpaliotis D, Alaswad K, Lombardi W, Grantham JA, Michael TT, Patel VG, Rangan BV, Kotsia AP, Lembo N, Kandzari DE, Lee J, Kalynych A, Carlson H, Garcia S, Banerjee S, Thompson CA, Brilakis ES. Application of the "hybrid approach" to chronic total occlusions in patients with previous coronary artery bypass graft surgery (from a Contemporary Multicenter US registry). Am J Cardiol. 2014 Jun 15;113(12):1990-4. doi: 10.1016/j.amjcard.2014.03.039. Epub 2014 Mar 31. PMID 24793678
- [Result] Christopoulos G, Karmpaliotis D, Alaswad K, Lombardi WL, Grantham JA, Rangan BV, Kotsia AP, Lembo N, Kandzari DE, Lee J, Kalynych A, Carlson H, Garcia S, Banerjee S, Thompson CA, Brilakis ES. The efficacy of "hybrid" percutaneous coronary intervention in chronic total occlusions caused by in-stent restenosis: insights from a US multicenter registry. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):646-51. doi: 10.1002/ccd.25465. Epub 2014 Jul 4. PMID 24585508
- [Result] Christopoulos G, Karmpaliotis D, Wyman MR, Alaswad K, McCabe J, Lombardi WL, Grantham JA, Marso SP, Kotsia AP, Rangan BV, Garcia SA, Lembo N, Kandzari D, Lee J, Kalynych A, Carlson H, Thompson CA, Banerjee S, Brilakis ES. Percutaneous intervention of circumflex chronic total occlusions is associated with worse procedural outcomes: insights from a Multicentre US Registry. Can J Cardiol. 2014 Dec;30(12):1588-94. doi: 10.1016/j.cjca.2014.07.007. Epub 2014 Jul 16. PMID 25442459
- [Result] Christopoulos G, Menon RV, Karmpaliotis D, Alaswad K, Lombardi W, Grantham A, Patel VG, Rangan BV, Kotsia AP, Lembo N, Kandzari D, Carlson H, Garcia S, Banerjee S, Thompson CA, Brilakis ES. The efficacy and safety of the "hybrid" approach to coronary chronic total occlusions: insights from a contemporary multicenter US registry and comparison with prior studies. J Invasive Cardiol. 2014 Sep;26(9):427-32. PMID 25198485
- [Result] Sapontis J, Christopoulos G, Grantham JA, Wyman RM, Alaswad K, Karmpaliotis D, Lombardi WL, McCabe JM, Marso SP, Kotsia AP, Rangan BV, Christakopoulos GE, Garcia S, Thompson CA, Banerjee S, Brilakis ES. Procedural failure of chronic total occlusion percutaneous coronary intervention: Insights from a multicenter US registry. Catheter Cardiovasc Interv. 2015 Jun;85(7):1115-22. doi: 10.1002/ccd.25807. Epub 2015 Feb 3. PMID 25557905
- [Result] Christopoulos G, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman RM, Lombardi WL, Menon RV, Grantham JA, Kandzari DE, Lembo N, Moses JW, Kirtane AJ, Parikh M, Green P, Finn M, Garcia S, Doing A, Patel M, Bahadorani J, Tarar MN, Christakopoulos GE, Thompson CA, Banerjee S, Brilakis ES. Application and outcomes of a hybrid approach to chronic total occlusion percutaneous coronary intervention in a contemporary multicenter US registry. Int J Cardiol. 2015 Nov 1;198:222-8. doi: 10.1016/j.ijcard.2015.06.093. Epub 2015 Jun 27. PMID 26189193
- [Result] Christopoulos G, Wyman RM, Alaswad K, Karmpaliotis D, Lombardi W, Grantham JA, Yeh RW, Jaffer FA, Cipher DJ, Rangan BV, Christakopoulos GE, Kypreos MA, Lembo N, Kandzari D, Garcia S, Thompson CA, Banerjee S, Brilakis ES. Clinical Utility of the Japan-Chronic Total Occlusion Score in Coronary Chronic Total Occlusion Interventions: Results from a Multicenter Registry. Circ Cardiovasc Interv. 2015 Jul;8(7):e002171. doi: 10.1161/CIRCINTERVENTIONS.114.002171. PMID 26162857
- [Result] Alaswad K, Menon RV, Christopoulos G, Lombardi WL, Karmpaliotis D, Grantham JA, Marso SP, Wyman MR, Pokala NR, Patel SM, Kotsia AP, Rangan BV, Lembo N, Kandzari D, Lee J, Kalynych A, Carlson H, Garcia SA, Thompson CA, Banerjee S, Brilakis ES. Transradial approach for coronary chronic total occlusion interventions: Insights from a contemporary multicenter registry. Catheter Cardiovasc Interv. 2015 Jun;85(7):1123-9. doi: 10.1002/ccd.25827. Epub 2015 Feb 3. PMID 25640902
- [Result] Danek BA, Karatasakis A, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Patel M, Bahadorani J, Lombardi WL, Wyman MR, Grantham JA, Doing A, Moses JW, Kirtane A, Parikh M, Ali ZA, Kalra S, Kandzari DE, Lembo N, Garcia S, Rangan BV, Thompson CA, Banerjee S, Brilakis ES. Use of antegrade dissection re-entry in coronary chronic total occlusion percutaneous coronary intervention in a contemporary multicenter registry. Int J Cardiol. 2016 Jul 1;214:428-37. doi: 10.1016/j.ijcard.2016.03.215. Epub 2016 Apr 6. PMID 27088405
- [Result] Karacsonyi J, Karatasakis A, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman MR, Lombardi WL, Grantham JA, Kandzari DE, Lembo N, Moses JW, Kirtane AJ, Parikh MA, Green P, Finn M, Garcia S, Doing A, Patel M, Bahadorani J, Martinez Parachini JR, Resendes E, Rangan BV, Ungi I, Thompson CA, Banerjee S, Brilakis ES. Effect of Previous Failure on Subsequent Procedural Outcomes of Chronic Total Occlusion Percutaneous Coronary Intervention (from a Contemporary Multicenter Registry). Am J Cardiol. 2016 Apr 15;117(8):1267-71. doi: 10.1016/j.amjcard.2016.01.021. Epub 2016 Jan 28. PMID 26899493
- [Result] Nguyen-Trong PK, Rangan BV, Karatasakis A, Danek BA, Christakopoulos GE, Martinez-Parachini JR, Resendes E, Ayers CR, Luna M, Abdullah S, Kumbhani DJ, Addo T, Grodin J, Banerjee S, Brilakis ES. Predictors and Outcomes of Side-Branch Occlusion in Coronary Chronic Total Occlusion Interventions. J Invasive Cardiol. 2016 Apr;28(4):168-73. Epub 2016 Jan 15. PMID 26773239
- [Result] Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, Alaswad K, Lombardi W, Grantham JA, Moses J, Christakopoulos G, Tarar MNJ, Rangan BV, Lembo N, Garcia S, Cipher D, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016 Jan 11;9(1):1-9. doi: 10.1016/j.jcin.2015.09.022. PMID 26762904
- [Result] Karatasakis A, Tarar MN, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman RM, Lombardi WL, Grantham JA, Kandzari DE, Lembo NJ, Moses JW, Kirtane AJ, Parikh M, Garcia S, Doing A, Pershad A, Shah A, Patel M, Bahadorani J, Shoultz CA Jr, Danek BA, Thompson CA, Banerjee S, Brilakis ES. Guidewire and microcatheter utilization patterns during antegrade wire escalation in chronic total occlusion percutaneous coronary intervention: Insights from a contemporary multicenter registry. Catheter Cardiovasc Interv. 2017 Mar 1;89(4):E90-E98. doi: 10.1002/ccd.26568. Epub 2016 May 17. PMID 27184465
- [Result] Christakopoulos GE, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman RM, Lombardi W, Grantham JA, Kandzari DA, Lembo N, Moses JW, Kirtane A, Parikh M, Green P, Finn M, Garcia S, Doing A, Patel M, Bahadorani J, Christopoulos G, Karatasakis A, Thompson CA, Banerjee S, Brilakis ES. Contrast Utilization During Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From a Contemporary Multicenter Registry. J Invasive Cardiol. 2016 Jul;28(7):288-94. PMID 27342206
- [Result] Nguyen-Trong PK, Alaswad K, Karmpaliotis D, Lombardi W, Grantham JA, Lembo N, Kandzari D, Karatasakis A, Karacsonyi J, Danek BA, Rangan BV, Roesle M, Ayers CR, Thompson CA, Banerjee S, Brilakis ES. Use of Saphenous Vein Bypass Grafts for Retrograde Recanalization of Coronary Chronic Total Occlusions: Insights From a Multicenter Registry. J Invasive Cardiol. 2016 Jun;28(6):218-24. PMID 27236005
- [Result] Danek BA, Karatasakis A, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel MP, Bahadorani J, Lombardi WL, Wyman RM, Grantham JA, Kandzari DE, Lembo NJ, Doing AH, Toma C, Moses JW, Kirtane AJ, Ali ZA, Parikh M, Garcia S, Nguyen-Trong PK, Karacsonyi J, Alame AJ, Kalsaria P, Thompson C, Banerjee S, Brilakis ES. Effect of Lesion Age on Outcomes of Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From a Contemporary US Multicenter Registry. Can J Cardiol. 2016 Dec;32(12):1433-1439. doi: 10.1016/j.cjca.2016.04.007. Epub 2016 Apr 22. PMID 27476986
- [Result] Karmpaliotis D, Karatasakis A, Alaswad K, Jaffer FA, Yeh RW, Wyman RM, Lombardi WL, Grantham JA, Kandzari DE, Lembo NJ, Doing A, Patel M, Bahadorani JN, Moses JW, Kirtane AJ, Parikh M, Ali ZA, Kalra S, Nguyen-Trong PK, Danek BA, Karacsonyi J, Rangan BV, Roesle MK, Thompson CA, Banerjee S, Brilakis ES. Outcomes With the Use of the Retrograde Approach for Coronary Chronic Total Occlusion Interventions in a Contemporary Multicenter US Registry. Circ Cardiovasc Interv. 2016 Jun;9(6):10.1161/CIRCINTERVENTIONS.115.003434 e003434. doi: 10.1161/CIRCINTERVENTIONS.115.003434. PMID 27307562
- [Result] Karatasakis A, Danek BA, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel MP, Bahadorani JN, Wyman RM, Lombardi WL, Grantham JA, Kandzari DE, Lembo NJ, Doing AH, Moses JW, Kirtane AJ, Garcia S, Parikh MA, Ali ZA, Karacsonyi J, Kalra S, Rangan BV, Kalsaria P, Thompson CA, Banerjee S, Brilakis ES. Impact of Proximal Cap Ambiguity on Outcomes of Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From a Multicenter US Registry. J Invasive Cardiol. 2016 Oct;28(10):391-396. PMID 27705889
- [Result] Karatasakis A, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel MP, Bahadorani JN, Lombardi WL, Wyman RM, Grantham JA, Kandzari DE, Lembo NJ, Doing AH, Toma C, Moses JW, Kirtane AJ, Ali Z, Parikh M, Garcia S, Danek BA, Karacsonyi J, Alame A, Kalsaria P, Thompson C, Banerjee S, Brilakis ES. Approaches to percutaneous coronary intervention of right coronary artery chronic total occlusions: insights from a multicentre US registry. EuroIntervention. 2016 Dec 10;12(11):e1326-e1335. doi: 10.4244/EIJ-D-16-00265. PMID 27934609
- [Result] Karacsonyi J, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Bahadorani J, Doing A, Ali ZA, Karatasakis A, Danek BA, Rangan BV, Alame AJ, Banerjee S, Brilakis ES. Prevalence, indications and management of balloon uncrossable chronic total occlusions: Insights from a contemporary multicenter US registry. Catheter Cardiovasc Interv. 2017 Jul;90(1):12-20. doi: 10.1002/ccd.26780. Epub 2016 Sep 21. PMID 27650935
- [Result] Karatasakis A, Danek BA, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Bahadorani JN, Lombardi WL, Wyman RM, Grantham JA, Kandzari DE, Lembo NJ, Doing AH, Toma C, Moses JW, Kirtane AJ, Parikh MA, Ali ZA, Garcia S, Kalsaria P, Karacsonyi J, Alame AJ, Thompson CA, Banerjee S, Brilakis ES. Comparison of various scores for predicting success of chronic total occlusion percutaneous coronary intervention. Int J Cardiol. 2016 Dec 1;224:50-56. doi: 10.1016/j.ijcard.2016.08.317. Epub 2016 Aug 23. PMID 27611917
- [Result] Martinez-Parachini JR, Karatasakis A, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Bahadorani J, Doing A, Nguyen-Trong PK, Danek BA, Karacsonyi J, Alame A, Rangan BV, Thompson CA, Banerjee S, Brilakis ES. Impact of diabetes mellitus on acute outcomes of percutaneous coronary intervention in chronic total occlusions: insights from a US multicentre registry. Diabet Med. 2017 Apr;34(4):558-562. doi: 10.1111/dme.13272. Epub 2016 Nov 3. PMID 27743404
- [Result] Karatasakis A, Iwnetu R, Danek BA, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Kandzari DE, Lembo NJ, Patel M, Mahmud E, Lombardi WL, Wyman RM, Grantham JA, Doing AH, Toma C, Choi JW, Uretsky BF, Moses JW, Kirtane AJ, Ali ZA, Parikh M, Karacsonyi J, Rangan BV, Thompson CA, Banerjee S, Brilakis ES. The Impact of Age and Sex on In-Hospital Outcomes of Chronic Total Occlusion Percutaneous Coronary Intervention. J Invasive Cardiol. 2017 Apr;29(4):116-122. Epub 2017 Jan 15. PMID 28089997
- [Result] Garcia S, Alraies MC, Karatasakis A, Yannopoulos D, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel MP, Bahadorani J, Karacsonyi J, Kalsaria P, Danek B, Banerjee S, Brilakis ES. Coronary artery spatial distribution of chronic total occlusions: Insights from a large US registry. Catheter Cardiovasc Interv. 2017 Jul;90(1):23-30. doi: 10.1002/ccd.26844. Epub 2016 Nov 10. PMID 27860111
- [Result] Christakopoulos GE, Christopoulos G, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman MR, Lombardi WL, Tarar MN, Grantham JA, Kandzari DE, Lembo N, Moses JW, Kirtane AJ, Parikh M, Green P, Finn M, Garcia S, Doing AH, Hatem R, Thompson CA, Banerjee S, Brilakis ES. Predictors of Excess Patient Radiation Exposure During Chronic Total Occlusion Coronary Intervention: Insights From a Contemporary Multicentre Registry. Can J Cardiol. 2017 Apr;33(4):478-484. doi: 10.1016/j.cjca.2016.11.002. Epub 2016 Nov 11. PMID 28169091
- [Derived] Mutlu D, Strepkos D, Ser OS, Carvalho PEP, Alexandrou M, Jalli S, Azzalini L, Ybarra L, Alaswad K, Jaffer FA, Davies R, Rangan BV, Sandoval Y, Nicholas Burke M, Gorgulu S, Brilakis ES; PROGRESS-CTO Investigators. Traditional Versus Dual Lumen Microcatheter-Assisted Parallel Wiring in Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From the PROGRESS-CTO Registry. Catheter Cardiovasc Interv. 2025 May;105(6):1493-1501. doi: 10.1002/ccd.31472. Epub 2025 Mar 10. PMID 40065565
- [Derived] Mutlu D, Strepkos D, Carvalho PE, Alexandrou M, Al-Ogaili A, Jalli S, Alaswad K, Jaffer FA, Davies R, Poommipanit P, Frizzel J, Elbarouni B, Khatri JJ, Gorgulu S, Goktekin O, Ozdemir R, Uluganyan M, ElGuindy A, Sadek Y, Ahmed Y, Basir MB, Raj L, Ybarra L, Murad B, Rangan BV, Mastrodemos OC, Azzalini L, Sandoval Y, Burke MN, Brilakis ES. Use of the Ostial Flash balloon in aorto-ostial chronic total occlusion percutaneous coronary intervention. J Invasive Cardiol. 2025 May;37(5). doi: 10.25270/jic/24.00263. PMID 39808454
- [Derived] Rempakos A, Alexandrou M, Mutlu D, Choi JW, Poommipanit P, Khatri JJ, Young L, Jefferson B, Gorgulu S, Jaffer FA, Chandwaney R, Davies R, Benton S, Alaswad K, Azzalini L, Kearney KE, Krestyaninov O, Khelimskii D, Dattilo P, Reddy N, Abi-Rafeh N, Elguindy A, Goktekin O, Rangan BV, Mastrodemos OC, Al-Ogaili A, Sandoval Y, Burke NM, Brilakis ES, Basir MB. Validation of the BCIS CHIP Score in chronic total occlusion percutaneous coronary intervention. Catheter Cardiovasc Interv. 2024 May;103(6):856-862. doi: 10.1002/ccd.31045. Epub 2024 Apr 17. PMID 38629740
- [Derived] Al-Ogaili A, Alexandrou M, Rempakos A, Mutlu D, Choi JW, Poommipanit P, Khatri JJ, Alaswad K, Basir MB, Chandwaney RH, Gorgulu S, ElGuindy AM, Elbarouni B, Jaber W, Rinfret S, Nicholson W, Jaffer FA, Aygul N, Azzalini L, Kearney KE, Frizzell J, Davies R, Goktekin O, Rangan BV, Mastrodemos OC, Sandoval Y, Nicholas Burke M, Brilakis ES. Retrograde chronic total occlusion percutaneous coronary intervention via ipsilateral collaterals. Catheter Cardiovasc Interv. 2024 May;103(6):863-872. doi: 10.1002/ccd.31019. Epub 2024 Apr 2. PMID 38563074
- [Derived] Rempakos A, Alexandrou M, Mutlu D, Choi JW, Poommipanit P, Khatri JJ, Young L, Dattilo P, Sadek Y, Davies R, Gorgulu S, Jaffer FA, Chandwaney R, Jefferson B, Elbarouni B, Azzalini L, Kearney KE, Alaswad K, Basir MB, Krestyaninov O, Khelimskii D, Aygul N, Abi-Rafeh N, Elguindy A, Goktekin O, Rangan BV, Mastrodemos OC, Al-Ogaili A, Sandoval Y, Burke MN, Brilakis ES, Kalyanasundaram A. Predictors of successful primary antegrade wiring in chronic total occlusion percutaneous coronary intervention. J Invasive Cardiol. 2024 Jun;36(6). doi: 10.25270/jic/23.00305. PMID 38446022
- [Derived] Mutlu D, Rempakos A, Alexandrou M, Al-Ogaili A, Rangan BV, Mastrodemos OC, Sandoval Y, Burke MN, Brilakis ES. Radiation dose during contemporary percutaneous coronary interventions for chronic total occlusion: insights from the PROGRESS-CTO registry. J Invasive Cardiol. 2024 Apr;36(4). doi: 10.25270/jic/23.00281. PMID 38412437
- [Derived] Simsek B, Rempakos A, Kostantinis S, Karacsonyi J, Rinfret S, Jaber W, Nicholson W, Gorgulu S, Alaswad K, Khatri J, Poommipanit P, Aygul N, Krestyanino O, Khelimskii D, Uretsky B, Goktekin O, Dattilo P, Potluri S, Al-Azizi K, Mastrodemos OC, Rangan BV, Allana SS, Sandoval Y, Burke MN, Brilakis ES. Frequency and outcomes of ad hoc chronic total occlusion percutaneous coronary intervention: insights from the progress-cto registry. J Invasive Cardiol. 2023 Jul;35(7):E329-E340. doi: 10.25270/jic/23.00070. PMID 37769619
- [Derived] Simsek B, Rempakos A, Kostantinis S, Karacsonyi J, Gorgulu S, Alaswad K, Choi JW, Jaffer FA, Doshi D, Poommipanit P, Aygul N, Krestyaninov O, Khelimskii D, Uretsky B, Davies R, Goktekin O, ElGuindy A, Jefferson BK, Patel TN, Patel M, Sheikh A, Karmpaliotis D, Potluri S, Al-Azizi K, Mastrodemos OC, Rangan BV, Allana SS, Sandoval Y, Burke MN, Brilakis ES. Periprocedural Mortality in Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From the PROGRESS-CTO Registry. Circ Cardiovasc Interv. 2023 Jun;16(6):e012977. doi: 10.1161/CIRCINTERVENTIONS.123.012977. Epub 2023 Jun 1. PMID 37259859
- [Derived] Simsek B, Khatri J, Young L, Kostantinis S, Karacsonyi J, Rempakos A, Alaswad K, Jaffer FA, Doshi D, Gorgulu S, Goktekin O, Kerrigan J, Haddad EV, Rinfret S, Jaber WA, Nicholson W, Krestyaninov O, Khelimskii D, Choi JW, Patel TN, Jefferson BK, Bradley SM, Rao SV, Rangan BV, Allana SS, Sandoval Y, Burke MN, Brilakis ES, Poommipanit PB; PROGRESS-CTO investigators. Same day discharge versus overnight observation following chronic total occlusion percutaneous coronary intervention: Insights from the PROGRESS-CTO registry. Catheter Cardiovasc Interv. 2023 May;101(6):1028-1035. doi: 10.1002/ccd.30644. Epub 2023 Mar 24. PMID 36960766
- [Derived] Simsek B, Kostantinis S, Karacsonyi J, Gorgulu S, Alaswad K, Jaffer FA, Doshi D, Khatri J, Poommipanit P, Aygul N, Abi Rafeh N, Krestyaninov O, Khelimskii D, Uretsky B, Davies R, Goktekin O, ElGuindy A, Jefferson BK, Patel TN, Patel M, Mastrodemos OC, Rangan BV, Allana S, Sandoval Y, Burke MN, Brilakis ES. Outcomes of Patients With Acute Coronary Syndromes Undergoing Chronic Total Occlusion Percutaneous Coronary Intervention. J Invasive Cardiol. 2023 Jan;35(1):E24-E30. doi: 10.25270/jic/22.00258. Epub 2022 Dec 15. PMID 36525540
- [Derived] Simsek B, Kostantinis S, Karacsonyi J, Alaswad K, Karmpaliotis D, Masoumi A, Jaffer FA, Doshi D, Khatri J, Poommipanit P, Gorgulu S, Abi Rafeh N, Goktekin O, Krestyaninov O, Davies R, ElGuindy A, Haddad EV, Kerrigan J, Patel M, Chandwaney RH, Mastrodemos OC, Allana S, Rangan BV, Brilakis ES. Predictors of success in primary retrograde strategy in chronic total occlusion percutaneous coronary intervention: insights from the PROGRESS-chronic total occlusion registry. Catheter Cardiovasc Interv. 2022 Jul;100(1):19-27. doi: 10.1002/ccd.30228. Epub 2022 May 26. PMID 35615875
- [Derived] Simsek B, Kostantinis S, Karacsonyi J, Alaswad K, Karmpaliotis D, Masoumi A, Jaffer FA, Doshi D, Khatri J, Poommipanit P, Gorgulu S, Abi Rafeh N, Goktekin O, Krestyaninov O, Davies R, ElGuindy A, Jefferson BK, Patel TN, Patel M, Chandwaney RH, Mastrodemos OC, Rangan BV, Brilakis ES. Prevalence and outcomes of balloon undilatable chronic total occlusions: Insights from the PROGRESS-CTO. Int J Cardiol. 2022 Sep 1;362:42-46. doi: 10.1016/j.ijcard.2022.04.057. Epub 2022 Apr 26. PMID 35483480
- [Derived] Vemmou E, Alaswad K, Khatri JJ, Nikolakopoulos I, Karacsonyi J, Xenogiannis I, Karmpaliotis D, Garcia S, Burke MN, Brilakis ES. Patient Radiation Dose During Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From the PROGRESS-CTO Registry. Circ Cardiovasc Interv. 2020 Oct;13(10):e009412. doi: 10.1161/CIRCINTERVENTIONS.120.009412. Epub 2020 Sep 25. No abstract available. PMID 32972204
- [Derived] Tajti P, Xenogiannis I, Gargoulas F, Karmpaliotis D, Alaswad K, Jaffer FA, Patel MP, Burke MN, Garcia S, Krestyaninov O, Koutouzis M, Jaber W, Brilakis ES; Collaborators. Technical and procedural outcomes of the retrograde approach to chronic total occlusion interventions. EuroIntervention. 2020 Dec 4;16(11):e891-e899. doi: 10.4244/EIJ-D-19-00441. PMID 31638578
- [Derived] Tajti P, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Mahmud E, Choi JW, Burke MN, Doing AH, Dattilo P, Toma C, Smith AJC, Uretsky B, Holper E, Potluri S, Wyman RM, Kandzari DE, Garcia S, Krestyaninov O, Khelimskii D, Koutouzis M, Tsiafoutis I, Jaber W, Samady H, Moses JW, Lembo NJ, Parikh M, Kirtane AJ, Ali ZA, Doshi D, Xenogiannis I, Stanberry LI, Rangan BV, Ungi I, Banerjee S, Brilakis ES. In-Hospital Outcomes of Chronic Total Occlusion Percutaneous Coronary Interventions in Patients With Prior Coronary Artery Bypass Graft Surgery. Circ Cardiovasc Interv. 2019 Mar;12(3):e007338. doi: 10.1161/CIRCINTERVENTIONS.118.007338. PMID 30871357
- [Derived] Tajti P, Alaswad K, Karmpaliotis D, Jaffer FA, Yeh RW, Patel M, Mahmud E, Choi JW, Burke MN, Doing AH, Dattilo P, Toma C, Smith AJC, Uretsky BF, Holper E, Potluri S, Wyman RM, Kandzari DE, Garcia S, Krestyaninov O, Khelimskii D, Koutouzis M, Tsiafoutis I, Khatri JJ, Jaber W, Samady H, Jefferson B, Patel T, Abdullah S, Moses JW, Lembo NJ, Parikh M, Kirtane AJ, Ali ZA, Doshi D, Xenogiannis I, Stanberry LI, Rangan BV, Ungi I, Banerjee S, Brilakis ES. Procedural Outcomes of Percutaneous Coronary Interventions for Chronic Total Occlusions Via the Radial Approach: Insights From an International Chronic Total Occlusion Registry. JACC Cardiovasc Interv. 2019 Feb 25;12(4):346-358. doi: 10.1016/j.jcin.2018.11.019. PMID 30784639
- [Derived] Tajti P, Burke MN, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Mahmud E, Choi JW, Doing AH, Datilo P, Toma C, Smith AJC, Uretsky B, Holper E, Garcia S, Krestyaninov O, Khelimskii D, Koutouzis M, Tsiafoutis I, Moses JW, Lembo NJ, Parikh M, Kirtane AJ, Ali ZA, Doshi D, Jaber W, Samady H, Rangan BV, Xenogiannis I, Ungi I, Banerjee S, Brilakis ES. Prevalence and Outcomes of Percutaneous Coronary Interventions for Ostial Chronic Total Occlusions: Insights From a Multicenter Chronic Total Occlusion Registry. Can J Cardiol. 2018 Oct;34(10):1264-1274. doi: 10.1016/j.cjca.2018.07.472. Epub 2018 Jul 31. PMID 30269827
- [Derived] Tajti P, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Mahmud E, Choi JW, Burke MN, Doing AH, Dattilo P, Toma C, Smith AJC, Uretsky B, Holper E, Wyman RM, Kandzari DE, Garcia S, Krestyaninov O, Khelimskii D, Koutouzis M, Tsiafoutis I, Moses JW, Lembo NJ, Parikh M, Kirtane AJ, Ali ZA, Doshi D, Rangan BV, Ungi I, Banerjee S, Brilakis ES. The Hybrid Approach to Chronic Total Occlusion Percutaneous Coronary Intervention: Update From the PROGRESS CTO Registry. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1325-1335. doi: 10.1016/j.jcin.2018.02.036. Epub 2018 Apr 26. PMID 29706508
- [Derived] Tajti P, Karmpaliotis D, Alaswad K, Toma C, Choi JW, Jaffer FA, Doing AH, Patel M, Mahmud E, Uretsky B, Karatasakis A, Karacsonyi J, Danek BA, Rangan BV, Banerjee S, Ungi I, Brilakis ES. Prevalence, Presentation and Treatment of 'Balloon Undilatable' Chronic Total Occlusions: Insights from a Multicenter US Registry. Catheter Cardiovasc Interv. 2018 Mar 1;91(4):657-666. doi: 10.1002/ccd.27510. Epub 2018 Jan 23. PMID 29359452
- [Derived] Danek BA, Karatasakis A, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Patel MP, Mahmud E, Lombardi WL, Wyman MR, Grantham JA, Doing A, Kandzari DE, Lembo NJ, Garcia S, Toma C, Moses JW, Kirtane AJ, Parikh MA, Ali ZA, Karacsonyi J, Rangan BV, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Scoring System for Predicting Periprocedural Complications During Percutaneous Coronary Interventions of Chronic Total Occlusions: The Prospective Global Registry for the Study of Chronic Total Occlusion Intervention (PROGRESS CTO) Complications Score. J Am Heart Assoc. 2016 Oct 11;5(10):e004272. doi: 10.1161/JAHA.116.004272. PMID 27729332
- [Derived] Karacsonyi J, Alaswad K, Jaffer FA, Yeh RW, Patel M, Bahadorani J, Karatasakis A, Danek BA, Doing A, Grantham JA, Karmpaliotis D, Moses JW, Kirtane A, Parikh M, Ali Z, Lombardi WL, Kandzari DE, Lembo N, Garcia S, Wyman MR, Alame A, Nguyen-Trong PK, Resendes E, Kalsaria P, Rangan BV, Ungi I, Thompson CA, Banerjee S, Brilakis ES. Use of Intravascular Imaging During Chronic Total Occlusion Percutaneous Coronary Intervention: Insights From a Contemporary Multicenter Registry. J Am Heart Assoc. 2016 Aug 20;5(8):e003890. doi: 10.1161/JAHA.116.003890. PMID 27543800
- See also: Official website of the Progress-CTO registry — http://www.progresscto.org/